CLINICAL TRIAL: NCT04516928
Title: Study of SARS-CoV2 Virus (COVID-19) Seroprevalence Among Lyon-Bron Military Health Schools Personnel
Acronym: SeroCovEms
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-29; 2020-A02125-34 (Other: IDRCB)
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: SARS-CoV Infection; Covid19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Anti-SARS-CoV2 Serology — The anti-SARS-CoV2 serological status will be measured on a blood sample collected at Day 0.
Other: Questionnaire — A questionnaire on socio-demographical status, health status and lifestyle habits during the pandemic will be filled by the participants at Day 0.

SUMMARY:
Emerging in China in December 2019, Covid-19, whose pathogen is SARS-Cov-2, was declared a global pandemic in March 2020. The clinical presentation is highly variable, ranging from asymptomatic forms to acute respiratory distress and even death. Transmission is by droplet route, with an R0 of approximately 3.

Rapidly, population protection measures were put in place by governments, including the confinement of all persons whose functions were not considered essential and the closure of educational institutions.

Health care institutions are places at risk of Covid-19 transmission and hospital staff are particularly exposed, either through direct contact with patients, contact with exposed persons or through the environment. In order to protect personnel, hygiene measures were immediately recalled and reinforced.

During the period of containment, the majority of students from the Lyon-Bron Military Medical Schools were sent as reinforcement in Army Training Hospitals and in the Military Reanimation Unit (Mulhouse). Some students developed symptomatic forms of SARS-Cov-2 infection, documented by positive PCR, during Operation Resilience or on their return from the mission.

The Lyon-Bron Military Medical Schools staff, exposed both to the initial phase of the epidemic and to national protection measures, represent an extremely interesting population for understanding the epidemiological dynamics of the virus.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* personnel of the Military Health Schools of Lyon-Bron
* working at the Military Health Schools of Lyon-Bron during the COVID-19 crisis

Exclusion Criteria:

* under 18
* contraindication to blood sampling

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of personnel of the Military Health Schools of Lyon-Bron (students, teachers, supervisors).
Sampling Method: Non-Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Proportion of anti-SARS-CoV2 seropositive participants | Day 0
  The proportion of anti-SARS-CoV2 seropositive participants will be determined. ELISA serology test will be used to detect anti-SARS-CoV2 antibodies (IgG and IgM) at Day 0.

SECONDARY OUTCOMES:
Proportion of asymptomatic participants (among anti-SARS-CoV2 seropositive participants) | Day 0
  The proportion of asymptomatic participants (among anti-SARS-CoV2 seropositive participants) will be determined. COVID-19 symptoms will be measured using a questionnaire.
Correlation coefficient between medical risk factors and a positive serology | Day 0
  Correlation coefficient between medical risk factors and a positive serology will be assessed using a step-by-step top-down regression analysis.
Correlation coefficient between epidemiological risk factors and a positive serology | Day 0
  Correlation coefficient between epidemiological risk factors and a positive serology will be assessed using a step-by-step top-down regression analysis.
Correlation coefficient between social risk factors and a positive serology | Day 0
  Correlation coefficient between social risk factors and a positive serology will be assessed using a step-by-step top-down regression analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Antenne Médicale des Ecoles Militaires de Santé de Lyon-Bron (EMSLB), Bron, France

IPD SHARING:
Plan to Share IPD: Undecided